CLINICAL TRIAL: NCT06274346
Title: Effect of Retro Walking Versus Isometric Multi-angular Exercises on Pain and Functional Performance in Knee Osteoarthritis in Geriatric Population: A Randomized Controlled Study
Brief Title: Effect of Retro Walking Versus Isometric Multi-angular Exercises on Pain and Functional Performance in Knee Osteoarthritis in Geriatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ahmedU
Record Dates: First submitted 2024-01-30; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned into two groups through computer software. We put sixty patients on the software program and the program assigned them randomly. s exercise, straight leg raise, prone knee bending, side lying hip abduction, prone hip extension with 5 seconds hold and a rest interval of 2 seconds for 10 repetitions for each exercise for a period of 4 weeks, 3 days per week was given. Second group was treated by retrowalking exercises in addition to physical therapy interventions including short wave diathermy and strengthening exercise such as static quadriceps exercise, dynamic quadriceps exercise, straight leg raise, prone knee bending, side lying hip abduction, prone hip extension with 5 seconds hold and a rest interval of 2 seconds for 10 repetitions for each exercise for a period of 4 weeks, 3 days per week was given., which were given 3 times/week for 4 consecutive weeks.
Who Masked: Participant
Masking Description: Sixty male and female geriatric patients had chronic knee osteoarthritis were chosen the outpatient clinic of faculty of physical therapy, Delta University for science and technology. education, occupation and duration of complaints of each patient. All were evaluated at the beginning of the treatment (week 0), at the endpoint of the treatment (week 4).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multiangular Isometric exercise group: (Active Comparator): Each patient was allowed to warm up for 10 minutes on the bicycle ergometer before each isometric exercise session. For this part of the study we position the patient on isokinetic device with the hip joint flexed at 90˚ the back supported with a backrest and the pelvis stabilized with a strap. The distal of the thigh was rested on a lifted support in the front of the seat and was wrapped with a strap. The center of rotation of the dynamometer was placed opposite the center of the femur lateral epicondyle. The lever arm of the dynamometer was set so that the load cell pad was comfortable against the lower part of the leg close to the lateral malleolus.
  Interventions: Other: Multiangular Isometric exercise
- Retrograde walking group: (Experimental): Each patient was allowed to warm up for 10 minutes on the bicycle ergometer before each retrograde walking session. The patients were instructed to walk backwards for 10 min on a flat surface for a distance of 30 m at a comfortable speed supervised by the physiotherapist. Patients were required to walk backwards without looking behind. Safety measures were taken to ensure patients' well-being during retro walking. The physiotherapist stood beside the patients, gave them moral support, and guided them through the walking path till the patients are confident to walk on their own. The patient is also encouraged to increase their speed throughout the 4 weeks of rehabilitation.
  Interventions: Other: Multiangular Isometric exercise
- Pulsed short wave diathermy: (Other): Patient is in supine lying, contra planer (transverse) method was used. The electrodes were placed over opposite aspects of the part i.e. knee. Timing: was applied for 20 minutes, 3 days/ week for duration of 4 weeks. After pulsed SWD, both groups were given static quadriceps exercise, dynamic quadriceps exercise, straight leg raise, prone knee bending, side lying hip abduction, prone hip extension for 10 repetitions with 5 seconds hold followed by 2 seconds rest for each exercise for a period of 3 days per week for duration of 4 weeks.
  Interventions: Other: Multiangular Isometric exercise

INTERVENTIONS:
Other: Multiangular Isometric exercise — already were described in arm descriptions
  Other Names: Retrograde walking

SUMMARY:
Osteoarthritis is a leading musculoskeletal cause of disability in elderly persons all over the world and a major cause of physical limitations and reduced quality of life (1). Its onset is around 40 years of age and it is estimated that over 80% of people over 55 have evidence of radiographic changes in the knee due to osteoarthritis. It has been estimated that the incidence has increased by the increase in life expectancy and it has been identified as a frequent cause for health services demand in patients over 65(2).

The common clinical manifestations of knee OA include pain, stiffness, joint enlargement, crepitus, muscle weakness, deformity, impaired proprioception, reduced joint motion, and disability(3).

Patients with knee Osteoarthritis seems to develop their own gait pattern and try to unload the affected structures during gait. More over patients with less severe knee osteoarthritis develop a gait pattern that differs from patients with severe osteoarthritis and control group of patients (4).

Isometric exercises are types of strength training in which the joint angle and muscle length do not change during contraction, and therefore this approach can be advantageous in the early stages of knee rehabilitation in cases where the range of motion is restricted due to pain (13). No physical work is performed during isometric exercise. Intensity and duration combination reflects the energy consumption of an isometric contraction (14). In addition, muscle strength increases in isometric exercise are specific to the angle applied. It was also concluded that isometric exercise performed at different angles should be especially considered as an alternative strength training since it induces the most noticeable and fastest increase in muscle moment (15). A study was conducted to investigate the effects of isometric quadriceps exercise on muscle strength, pain, and function in knee osteoarthritis, it was concluded that isometric quadriceps exercise program showed beneficial effects on quadriceps muscle strength, pain, and functional disability in patients with osteoarthritis of the knee (16).

Another study was conducted to assess the effectiveness of Isometric exercise and counseling on level of pain among patients with Knee osteoarthritis, the authors concluded that Isometric exercise and counseling program has significantly reduced pain, stiffness and improved physical function and the authors recommended that Isometric exercise and counselling should be adopted as a routine care in the hospitals treating patients with knee osteoarthritis (17) Thus, we hypothesized that a less intensive walking program such as retro walking program could provide an additional benefit more than those experienced by forward walking program in the previous studies. Therefore, the primary aim of the present study was to compare the effect of retro walking versus isometric multiangular exercises group on knee pain and function in geriatric people.

Materials and Methods

This randomized controlled experimental trial was carried out at the outpatient clinic of faculty of physical therapy, Delta University for science and technology from June 2023 to November 2023. The aims of the study and the study protocol were explained for each patient before participation in the study. All patients signed an approved informed consent form for participation in this study. Before starting the treatment program, a complete history and physical examination will be taken for all patients.

Subjects:

Sixty male and female geriatric patients had chronic knee osteoarthritis were chosen the outpatient clinic of faculty of physical therapy, Delta University for science and technology. In each case, the diagnosis of knee OA was based on the criteria specified by the American College of Rheumatology.

We recorded the height, weight, and medical history, and lower extremity dominance, level of education, occupation and duration of complaints of each patient. All were evaluated at the beginning of the treatment (week 0), at the endpoint of the treatment (week 4)

DETAILED DESCRIPTION:
Introduction:

Osteoarthritis is a leading musculoskeletal cause of disability in elderly persons all over the world and a major cause of physical limitations and reduced quality of life (1). Its onset is around 40 years of age and it is estimated that over 80% of people over 55 have evidence of radiographic changes in the knee due to osteoarthritis. It has been estimated that the incidence has increased by the increase in life expectancy and it has been identified as a frequent cause for health services demand in patients over 65(2).

The common clinical manifestations of knee OA include pain, stiffness, joint enlargement, crepitus, muscle weakness, deformity, impaired proprioception, reduced joint motion, and disability(3).

Patients with knee Osteoarthritis seems to develop their own gait pattern and try to unload the affected structures during gait. More over patients with less severe knee osteoarthritis develop a gait pattern that differs from patients with severe osteoarthritis and control group of patients (4).

Biomechanical studies indicated individual with O.A. knee walk more slowly, with less knee excursion, increased adduction moment and with more joint stiffness. These secondary compensatory gait adaptation in O.A. knee patients helps in reducing pain by decreasing ground reaction loading on knee (5). This prolonged usage of secondary gait compensation creates greater imbalances of muscle, progressively reduces muscle strength, endurance, flexibility and later ending to deformity (6).

Therapeutic exercises are often used to improve physiological impairments such as reduced joint motion, muscle weakness, impaired balance, disability, and proprioception(7).

Retro-walking is sometimes referred to as backward walking, has been thought to be used already for several decades in China, Japan and Europe to get a physical workout, improve sport performance, promote balance and also to stay mentally fit (8). Retro-walking is walking backwards (9).

Since there is propulsion in backward direction and reversal of leg movement in Retro-walking, different muscle activation patterns from those in forward walking are required (10). Backward walking increases stride rate, decreases stride length and increases support time. Muscular structure supporting ankle and knee reversed their role during retro-walking. Backward walking produces significantly lower patellar compressive force than forward walking and helps to reduce maximal vertical force and impulsive force on knee in comparison to forward walking because of Toe heel contact pattern. Retro-walking is associated with increased cadence, decreased stride length and different joint kinematics as compared to forward walking and hence may offer some benefits over forward walking alone (11, 12).

Isometric exercises are types of strength training in which the joint angle and muscle length do not change during contraction, and therefore this approach can be advantageous in the early stages of knee rehabilitation in cases where the range of motion is restricted due to pain (13). No physical work is performed during isometric exercise. Intensity and duration combination reflects the energy consumption of an isometric contraction (14). In addition, muscle strength increases in isometric exercise are specific to the angle applied. It was also concluded that isometric exercise performed at different angles should be especially considered as an alternative strength training since it induces the most noticeable and fastest increase in muscle moment (15). A study was conducted to investigate the effects of isometric quadriceps exercise on muscle strength, pain, and function in knee osteoarthritis, it was concluded that isometric quadriceps exercise program showed beneficial effects on quadriceps muscle strength, pain, and functional disability in patients with osteoarthritis of the knee (16).

Another study was conducted to assess the effectiveness of Isometric exercise and counseling on level of pain among patients with Knee osteoarthritis, the authors concluded that Isometric exercise and counseling program has significantly reduced pain, stiffness and improved physical function and the authors recommended that Isometric exercise and counselling should be adopted as a routine care in the hospitals treating patients with knee osteoarthritis (17) Thus, we hypothesized that a less intensive walking program such as retro walking program could provide an additional benefit more than those experienced by forward walking program in the previous studies. Therefore, the primary aim of the present study was to compare the effect of retro walking versus isometric multiangular exercises group on knee pain and function in geriatric people.

Materials and Methods

This randomized controlled experimental trial was carried out at the outpatient clinic of faculty of physical therapy, Delta University for science and technology from June 2023 to November 2023. The aims of the study and the study protocol were explained for each patient before participation in the study. All patients signed an approved informed consent form for participation in this study. Before starting the treatment program, a complete history and physical examination will be taken for all patients.

Subjects:

Sixty male and female geriatric patients had chronic knee osteoarthritis were chosen the outpatient clinic of faculty of physical therapy, Delta University for science and technology. In each case, the diagnosis of knee OA was based on the criteria specified by the American College of Rheumatology.

We recorded the height, weight, and medical history, and lower extremity dominance, level of education, occupation and duration of complaints of each patient. All were evaluated at the beginning of the treatment (week 0), at the endpoint of the treatment (week 4).

Inclusion criteria: Male and female geriatric participants clinically diagnosed with osteoarthritis of knee by Orthopaedician; Age more than 60 years; Participants having grade 2 and grade 3 as per Kellgren and Lawrence scale; The participants fulfilling clinical criteria listed by the American College of Rheumatology: knee pain and any three out of six: age > 50 years, morning stiffness lasting < 30 minutes, crepitus on active motion, bony tenderness, bony enlargement, no warmth on touch; Participants having knee pain for more than 6 weeks; Willingness to participate in the study.

Exclusion criteria: Participants with inflammatory joint disease of lower extremity, neurological disorder (motor and sensory loss), cardiac or metabolic condition; Participants involved in any form of physical exercise for lower extremity for at least 3 months; Participants taking pharmacological interventions; Participants taking an intra- articular injection for knee since last 6 months; Participants with history of recent surgery to hip, knee, ankle joint involving ligament, meniscus; Participants with balance problem.

Patients were randomly assigned into two groups through computer software. We put sixty patients on the software program and the program assigned them randomly. The first group was treated by isometric multiangular exercises in addition to physical therapy interventions including short wave diathermy and strengthening exercise such as static quadriceps exercise, dynamic quadriceps exercise, straight leg raise, prone knee bending, side lying hip abduction, prone hip extension with 5 seconds hold and a rest interval of 2 seconds for 10 repetitions for each exercise for a period of 4 weeks, 3 days per week was given. Second group was treated by retrowalking exercises in addition to physical therapy interventions including short wave diathermy and strengthening exercise such as static quadriceps exercise, dynamic quadriceps exercise, straight leg raise, prone knee bending, side lying hip abduction, prone hip extension with 5 seconds hold and a rest interval of 2 seconds for 10 repetitions for each exercise for a period of 4 weeks, 3 days per week was given., which were given 3 times/week for 4 consecutive weeks.

Procedures The patients were assessed twice; the first time was before the sessions. The second was at the end of the sessions. The visual analogue scale and the Western Ontario and McMaster Universities Arthritis Index (WOMAC) were examined by a physical therapist who was trained for all assessments for 10 days before this study and was blinded for the study objectives.

Assessment Pain intensity It was examined by using a 10 cm long visual analogue scale (VAS) during both rest and activity (0 = no pain, 10 = very severe pain).

Functional assessment:

It was assessed with the Western Ontario and McMaster Universities Arthritis Index (WOMAC), which consists of 24 questions, specifically 5 for pain, 2 for joint stiffness and 17 related to functional status, each being scored from 1 to 5 On this metric, a high score suggests bad health, while relatively healthy subjects will have a low score. The assessments were grouped into four classifications, specifically WOMAC A for pain, WOMAC B for joint stiffness, WOMAC C for function status, and WOMAC-Total for the total score.

Intervention procedures:

Multiangular Isometric exercise group:

Each patient was allowed to warm up for 10 minutes on the bicycle ergometer before each isometric exercise session. For this part of the study we position the patient on isokinetic device with the hip joint flexed at 90˚ the back supported with a backrest and the pelvis stabilized with a strap. The distal of the thigh was rested on a lifted support in the front of the seat and was wrapped with a strap. The center of rotation of the dynamometer was placed opposite the center of the femur lateral epicondyle. The lever arm of the dynamometer was set so that the load cell pad was comfortable against the lower part of the leg close to the lateral malleolus.

The patients were then positioned into the isokinetic test and exercise system as described previously. The angle of the knee joint is 0˚ when it is straight. Likewise, the isometric exercise programme was performed for affected knee 3 sessions a week for 4 weeks (12 sessions) on the isokinetic device. This system allowed us to perform isometric exercises at different angles. In this way, each knee of the patient was subject to 3 repetitions with maximum effort for 5 sec of isometric contraction to the knee flexor and extensor muscles at 0, 30, 45, and 60_ joint angles, with angular velocity 0˚/SEC and rest periods of 5 sec between each contraction, and rest periods of 30 sec at the change of each angle. (18)

Retrograde walking group:

Each patient was allowed to warm up for 10 minutes on the bicycle ergometer before each retrograde walking session. The patients were instructed to walk backwards for 10 min on a flat surface for a distance of 30 m at a comfortable speed supervised by the physiotherapist. Patients were required to walk backwards without looking behind. Safety measures were taken to ensure patients' well-being during retro walking. The physiotherapist stood beside the patients, gave them moral support, and guided them through the walking path till the patients are confident to walk on their own. The patient is also encouraged to increase their speed throughout the 4 weeks of rehabilitation. (19)

Pulsed short wave diathermy:

Patient is in supine lying, contra planer (transverse) method was used. The electrodes were placed over opposite aspects of the part i.e. knee. Timing: was applied for 20 minutes, 3 days/ week for duration of 4 weeks. After pulsed SWD, both groups were given static quadriceps exercise, dynamic quadriceps exercise, straight leg raise, prone knee bending, side lying hip abduction, prone hip extension for 10 repetitions with 5 seconds hold followed by 2 seconds rest for each exercise for a period of 3 days per week for duration of 4 weeks. (20)

ELIGIBILITY:
Inclusion Criteria:

* Male and female geriatric participants clinically diagnosed with osteoarthritis of knee by Orthopaedician; - Age more than 60 years
* Participants having grade 2 and grade 3 as per Kellgren and Lawrence scale
* The participants fulfilling clinical criteria listed by the American College of Rheumatology: knee pain and any three out of six: age > 50 years, morning stiffness lasting < 30 minutes, crepitus on active motion, bony tenderness, bony enlargement, no warmth on touch
* Participants having knee pain for more than 6 weeks; Willingness to participate in the study.

Exclusion Criteria:

* Participants with inflammatory joint disease of lower extremity, neurological disorder (motor and sensory loss), cardiac or metabolic condition
* Participants involved in any form of physical exercise for lower extremity for at least 3 months
* Participants taking pharmacological interventions
* Participants taking an intra- articular injection for knee since last 6 months
* Participants with history of recent surgery to hip, knee, ankle joint involving ligament, meniscus;
* Participants with balance problem

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | pre the intervention and immediately after the intervention
  It was examined by using a 10 cm long visual analogue scale (VAS) during both rest and activity (0 = no pain, 10 = very severe pain).
Functional assessment: | pre the intervention and immediately after the intervention
  It was assessed with the Western Ontario and McMaster Universities Arthritis Index (WOMAC), which consists of 24 questions, specifically 5 for pain, 2 for joint stiffness and 17 related to functional status, each being scored from 1 to 5 On this metric, a high score suggests bad health, while relatively healthy subjects will have a low score. The assessments were grouped into four classifications, specifically WOMAC A for pain, WOMAC B for joint stiffness, WOMAC C for function status, and WOMAC-Total for the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Delta University For Science and Technology, Gamasa, Almansourah, Egypt

IPD SHARING:
Plan to Share IPD: No